CLINICAL TRIAL: NCT01802177
Title: Efficacy and Safety of UVB Excimer Light in Alopecia Areata: A Prospective, Single-Blind Randomized Controlled Trial
Brief Title: Excimer Light for Alopecia Areata
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H12-02840
Record Dates: First submitted 2013-02-20; First posted 2013-03-01 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata; Excimer; UVB
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UVB excimer light (Experimental): Patches of alopecia will be treated twice weekly with UVB excimer light. Only one half of a single alopecia areata patch will be treated. In order to treat the same half during each visit, a transparent sheet will be marked, using a marking pen, to delineate the borders of the treatment area with a central dividing line. The other half will be covered and used as a control. Treatments will be given randomly (by sealed envelope randomization method) into one of the two halves in different patients but will be given into the same half in each patient in all treatment sessions. Only one investigator will know the intervention each half has received. A total of 23 treatments will be given over 12 weeks.
  Interventions: Procedure: UVB excimer light
- No treatment (covered) (No Intervention)

INTERVENTIONS:
Procedure: UVB excimer light
  Arms: UVB excimer light

SUMMARY:
Alopecia Areata (AA) is a chronic autoimmune inflammatory disease causing nonscarring hair loss. Many treatment modalities have been found to be helpful in AA, however, none on them cure the disease. UVB excimer light has recently emerged as a new therapeutic modality in many dermatologic diseases. There are no prospective randomized controlled trials evaluating the efficacy and safety of UVB excimer light in AA. We plan on conducting a prospective split lesion single-blinded randomized clinical trial to assess efficacy and safety of UVB excimer light in the treatment of AA.

DETAILED DESCRIPTION:
Alopecia Areata (AA) is a chronic autoimmune inflammatory disease causing nonscarring hair loss. Many treatment modalities have been found to be helpful in AA, however, none on them cure the disease.

Excimer laser has been shown to be effective in the treatment of AA in controlled studies. The main disadvantage of the previous studies evaluating excimer laser is choosing separate patches as a control which does not account for interlesional treatment response variability. UVB excimer light has recently emerged as a new therapeutic modality in many dermatologic diseases. However, there are only a few studies that evaluated the efficacy and safety of UVB excimer light in AA. Those studies have shown that UVB excimer light is effective in the treatment of AA but none of them was conducted in a controlled fashion.

There are no prospective randomized controlled trials evaluating the efficacy and safety of UVB excimer light in AA. We plan on conducting a prospective split lesion single-blinded randomized clinical trial to assess efficacy and safety of UVB excimer light in the treatment of AA.

Study Objectives

1. To evaluate the potential for UVB excimer light to induce hair regrowth within AA patches.
2. To assess the side effect profile of UVB excimer light when used in the treatment of AA.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Subject has a patch of at least 12 cm2 on the scalp with no evidence of hair regrowth.
* Subject is willing and capable of cooperating to the extent and degree required by the protocol.

Exclusion Criteria:

* Patients who received treatment for alopecia areata within the past 4 weeks.
* Patients with alopecia totalis or alopecia universalis.
* Patients with known photosensitivity like having polymorphous light eruption, connective tissue diseases, porphyria or Xeroderma pigmentosum.
* Pregnancy or breast-feeding.
* History of previous skin cancer.
* Patients that have participated in another investigational drug or device study within 30 days of enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of hair regrowth for each half. We will consider the treamtment successful if there was ≥50% hair regrowth from baseline. | at 6, 12, and 16 weeks from baseline

SECONDARY OUTCOMES:
Change in hair count and caliber in each half | at 6, 12, and 16 weeks from baseline
Assessment of side effects in each half | at 6, 12, and 16 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Lui, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- The Skin Care Center, Vancouver General Hospital, Vancouver, British Columbia, Canada